CLINICAL TRIAL: NCT05262725
Title: A Pilot Study of Behavioral Activation for People With Opioid Use Disorder
Brief Title: Behavioral Activation for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMCH-2022-30580
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; behavioral activation; primary care; buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: single-arm, pre/post pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Values-based Behavioral Activation (BA) (Experimental)
  Interventions: Behavioral: Values-based Behavioral Activation

INTERVENTIONS:
Behavioral: Values-based Behavioral Activation — Initially, patients complete a values assessment in which they identify personal values in various life domains. With the assistance of a clinician, patients set incremental behavior goals to move their daily actions to better align with their self-reported values. Goal completion allows the patient to achieve outcomes consistent with recovery, and they potentially experience enjoyment, self-efficacy, and confidence as they progress through the treatment.

SUMMARY:
The overall purpose of this pilot study is to evaluate the feasibility and acceptability of values-based behavioral activation (BA) as an adjunct intervention for patients receiving medications for opioid use disorder (OUD) in primary care. Researcher will evaluate the following aims: 1) examine the feasibility of BA for OUD in primary care, 2) examine whether the BA intervention and study requirements are acceptable to participants, and 3) determine the psychometric properties of the outcome measures in people with OUD. Participants will complete 4-6 brief counseling sessions over the course of 12 weeks. During the first session, participants will discuss values and recovery outcomes important to them. Next, they will set 2-3 personal goals to work on before the next BA session. At the follow-up sessions, participants will update the counselor on progress made or challenges experienced. Personal values will be reviewed and participant goals updated. Study measures (surveys and urine drug tests) will be completed at the start, partway through, and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Diagnosis of opioid use disorder.
* Have an active prescription for buprenorphine-naloxone (Suboxone) for at least one month.
* Patient at Broadway Family Medicine (BFM)

Exclusion Criteria:

* Concurrent individual psychotherapy with a psychologist or counselor at least monthly
* Active suicidal ideation (intention, plan, or attempt in the past 30 days, as determined by chart review)
* Dementia, developmental disabilities, or cognitive functioning that is too low to participate in therapy, as determined by chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment | 3 months from baseline
  % of patients approached who consent
Recruitment Pace | 3 months following intervention
  Average # of patients enrolled per week
Retention Percent | 3 months following intervention
  % of consented patients who complete the study
Treatment Satisfaction | 3 months following intervention
  Average satisfaction score

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levy, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Hooker SA, Kim H, Lonergan-Cullum M, Busch AM, Nissly T, Levy R. Adapting behavioral activation for patients receiving medications for opioid use disorder in primary care: a pilot study. Front Psychol. 2024 Oct 8;15:1439946. doi: 10.3389/fpsyg.2024.1439946. eCollection 2024. PMID 39439755

DOCUMENTS (1):
  • Informed Consent Form (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT05262725/ICF_000.pdf